CLINICAL TRIAL: NCT05562856
Title: Clinical Evaluation of White Spot Lesions Treated by Surface Pre-reacted Glass Filler Coating Material and Composite Sealants in Comparison With Icon Resin Infiltration by Using Laser Fluorescence and Spectrophotometer
Brief Title: Clinical Evaluation of White Spot Lesions Treated by S-PRG Material and Composite Sealants in Comparison With ICON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Eslam Gabr, Assistant professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 350/466/08/10/19
Record Dates: First submitted 2022-09-16; First posted 2022-10-03 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: White Spot Lesions

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- surface pre-reacted glass filler coating material (Experimental): surface pre-reacted glass filler coating material used to remineralize WSLs
  Interventions: Combination Product: surface pre-reacted glass filler coating material
- micro-invasive resin infiltration technique (Icon) (Active Comparator): micro-invasive resin infiltration technique (Icon) in the ability to improve caries lesion state (LF scores) and making the WSLs
  Interventions: Combination Product: surface pre-reacted glass filler coating material
- Permaseal resin (Experimental): Permaseal composite resin sealant as micro-invasive resin infiltration technique in the ability to improve caries lesion state (LF scores) and making the WSLs
  Interventions: Combination Product: surface pre-reacted glass filler coating material
- Optiguard resin (Experimental): Optiguardcomposite resin sealant as micro-invasive resin infiltration technique in the ability to improve caries lesion state (LF scores) and making the WSLs
  Interventions: Combination Product: surface pre-reacted glass filler coating material

INTERVENTIONS:
Combination Product: surface pre-reacted glass filler coating material — the ability to improve the aesthetic appearance (masking) and caries lesion state of the WSLs

SUMMARY:
Dental caries is the primary cause of tooth loss and oral diseases. Dental decay is a continuous pathological process with loss of tooth minerals, demineralization, which involves the destruction of tooth structure from acids. The first sign of early active demineralization is white spot lesions (WSLs) on the tooth surface, meanwhile, subsurface active mineral decomposition.

DETAILED DESCRIPTION:
Deposition of minerals depends on the equilibrium between demineralization and remineralization which may happen as a natural repair mechanism. The aim of this trial is to comparatively evaluate the efficacy of surface pre-reacted glass filler (S-PRG) Barrier Coat coating material against the Icon resin infiltration in the ability to improve the caries lesion state of the WSLs along 1 year. Laser fluorescence was used to compare the two materials to evaluate the caries progression. PRG Barrier Coat group showed immediate significant improvement in LF scores in demineralization progress and inhibition of caries progression with a significant improved effect. S-PRG Barrier Coat was clinically successful strategy in inhibition of caries and improve remineralization.

ELIGIBILITY:
Inclusion Criteria:

* Patients within 20-40 years of age.
* Each patient has 4 or more WSLs.
* Mild and moderate WSLs according to Gorelick's scale.
* Good oral hygiene and willing patients who can attend the study visits.
* a Symmetrical number of permanent teeth in each arch (mesial to second molars).

Exclusion Criteria:

* Active carious lesions.
* Facial surface restorations.
* Intrinsic and extrinsic stains.
* Patients who have a significant medical history or if they smoke.
* Criteria for discontinuation; Mortality and acquiring severe debilitating disease

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2021-12-02 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Assessments of caries lesion state of WSLs: | 1 year
  Assessing of carious lesions state of WSLs, was performed by using Diagnodent pen to record the progression or regression of caries by time. The assessment of the WSLs demineralization condition took place before intervention (baseline) [T0], immediately after intervention [T1], 3 months later [T2] ,6 months later [T3] and 1 year later [T4].

SECONDARY OUTCOMES:
Assessment of color change of WSLs: | 1 year
  The difference in color of the WSLs were performed by Vita Easyshade V at the five distinct times: before intervention (baseline) [T0], immediately after intervention [T1], 3 months later [T2] ,6 months later [T3] and 1 year later [T4].

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Noman, PROF, Study Director — Alazhar Univerisity
Locations (1):
- Mohamed Wakwak, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No